CLINICAL TRIAL: NCT01084707
Title: Multiple-dose Nicotine Pharmacokinetics With a New Oral Nicotine Replacement Product. A Study in Healthy Smokers.
Brief Title: Multiple-dose Nicotine Pharmacokinetics With a New Oral Nicotine Replacement Product.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NICTDP1066-A6431117; 2008-006279-65 (EudraCT Number)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Results first posted 2010-10-19 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Tobacco Dependence
Keywords: Smoking Cessation, Nicotine pharmacokinetics
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Nicotine; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Oral Nicotine 24-SA (Experimental): 2 Self-administrations of Experimental Nicotine once every hour
  Interventions: Drug: Oral Nicotine
- Oral Nicotine 24 (Experimental): 2 administrations of Experimental Nicotine by study personnel once every hour
  Interventions: Drug: Oral Nicotine
- Oral Nicotine 48 (Experimental): 2 administrations of Experimental Nicotine by study personnel once every 30 minutes
  Interventions: Drug: Oral Nicotine
- NiQuitin™ Lozenge 4 mg (Active Comparator): 1 NiQuitin™ lozenge, administered by study personnel once every hour
  Interventions: Drug: Nicotine Lozenge
- Nicorette® Gum 4 mg (Active Comparator): 1 piece Nicorette® gum, chewed for 30 minutes once every hour
  Interventions: Drug: Nicotine gum

INTERVENTIONS:
Drug: Oral Nicotine — Oral Nicotine either self-administered or provided by study personnel within 12 hours
  Other Names: generic Nicotine
  Arms: Oral Nicotine 24; Oral Nicotine 24-SA; Oral Nicotine 48
Drug: Nicotine Lozenge — Nicotine lozenge marketed as NiQuitin™ 4 mg hourly within 12 hours
  Other Names: NiQuitin™
  Arms: NiQuitin™ Lozenge 4 mg
Drug: Nicotine gum — Nicotine gum marketed as Nicorette® 4 mg hourly within 12 hours
  Other Names: Nicorette®
  Arms: Nicorette® Gum 4 mg

SUMMARY:
A comparison of three products for oral nicotine replacement with respect to pharmacokinetics after multiple-doses of nicotine.

DETAILED DESCRIPTION:
This study compares a new oral Nicotine Replacement Therapy (NRT) product with NiQuitin™ lozenge 4 mg and Nicorette®gum 4 mg, after 12 hours of nicotine abstinence, with respect to steady-state nicotine pharmacokinetics, during 12 hours after start of the first administration. Multiple doses of each treatment are given once hourly during five separate treatment visits scheduled in a crossover setting with randomized treatment sequences. The study will include 40 healthy smokers between 18-50 years, who have been smoking at least 20 cigarettes daily during at least one year preceding inclusion. Subjects and study personnel will be aware of which treatment is administered at a given visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy smokers, smoking at least 20 cigarettes daily during at least one year preceding inclusion and BMI between 17.5 and 30.0 kg/m2.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Treatment with an investigational product or donation or loss of blood within 3 month preceding the first dose of study medication.
* Prior regular use of nicotine mouth spray

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Clinical Pharmacology, Lund, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a five-arm cross-over trial, with subjects randomized to the order they received the different treatments and with analysis performed on valid pharmacokinetic data. Therefore, Number of Participants Analyzed in each arm represents the same subjects, and the total is not consistent with numbers provided in the participant flow module.
Groups:
- Overall Study: All subjects randomized into the trial
Period: Overall Study
Arm/Group | Overall Study
Started | 40
Completed | 34
Not Completed | 6
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Subjects: All subjects randomized into the trial, e.g., Full Analysis Set
Arm/Group | All Randomized Subjects
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 22
Region of Enrollment [Number; unit: participants]
  Sweden | 40

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration
Description: Cmax, which is the maximum (peak) concentration (amount of drug) measurable in blood plasma after a dose is administered measured in nanograms/milliliter (ng/ml)
Time Frame: During the last dosing interval (hour 11-12 post-dose)
Measure: Geometric Mean (Standard Deviation); unit: (ng/ml)
Groups:
- Oral Nicotine 24-SA: Oral Nicotine 24 mg, 2 1mg self-administrations once every hour; 12 doses of 2 mg over 11 hours
- Oral Nicotine 24: Oral Nicotine 24 mg, 2 1mg administrations by study personnel once every hour; 12 doses of 2 mg over 11 hours
- Oral Nicotine 48: Oral Nicotine 48 mg, 2 1mg administrations by study personnel once every 30 minutes; 24 doses of 2 mg over 11.5 hours
- NiQuitin™ Lozenge 4 mg: NiQuitin™ lozenge 4 mg; 12 doses of NiQuitin™ lozenge 4 mg over 11 hours
- Nicorette® Gum 4 mg: 12 doses of NICORETTE® gum 4 mg over 11 hours
Arm/Group | Oral Nicotine 24-SA | Oral Nicotine 24 | Oral Nicotine 48 | NiQuitin™ Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 39 | 35 | 32 | 35 | 32
(ng/ml) | 15.43 (6.12) | 16.49 (4.99) | 30.07 (9.77) | 27.07 (10.95) | 25.96 (8.55)

2. Secondary Outcome: Time of Maximum Concentration
Description: The time at which maximum concentration is reached (Tmax)
Time Frame: During the last dosing interval (hour 11-12 post-dose)
Population: ITT
Measure: Median (Full Range); unit: (minutes)
Arm/Group | Oral Nicotine 24-SA | Oral Nicotine 24 | Oral Nicotine 48 | NiQuitin™ Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 39 | 35 | 32 | 35 | 32
(minutes) | 15.0 (9.0) [5.0 to 42.0] | 10.0 (9.2) [5.0 to 45.0] | 10.0 (5.3) [5.0 to 23.0] | 25.0 (10.4) [13.0 to 55.0] | 30.0 (9.1) [10.0 to 50.0]

3. Secondary Outcome: Minimum Plasma Concentration
Description: The minimum nicotine plasma concentration during the last dosing interval (Cmin)
Time Frame: During the last dosing interval (hour 11-12 post-dose)
Population: ITT
Measure: Mean (Standard Deviation); unit: (ng/ml)
Arm/Group | Oral Nicotine 24-SA | Oral Nicotine 24 | Oral Nicotine 48 | NiQuitin™ Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 39 | 35 | 32 | 35 | 32
(ng/ml) | 11.54 (4.71) | 11.67 (4.04) | 25.32 (8.41) | 22.14 (9.71) | 19.00 (7.00)

4. Secondary Outcome: Peak-Trough Fluctuation
Description: Percent of peak-trough fluctuation over one dosing interval at steady state (PTF)
Time Frame: During the last dosing interval (hour 11-12 post-dose)
Population: ITT
Measure: Mean (Standard Deviation); unit: Percent Fluctuation
Arm/Group | Oral Nicotine 24-SA | Oral Nicotine 24 | Oral Nicotine 48 | NiQuitin™ Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 39 | 35 | 32 | 35 | 32
Percent Fluctuation | 35.6 (14.2) | 38.4 (14.9) | 21.7 (8.7) | 29.1 (10.7) | 36.3 (12.8)

5. Secondary Outcome: Nicotine Plasma Concentration
Description: The nicotine concentration in plasma (area under the nicotine plasma concentration curve) 1 hour after start of treatment
Time Frame: One hour after start of treatment
Population: ITT
Measure: Geometric Mean (Standard Deviation); unit: (ng/ml)
Arm/Group | Oral Nicotine 24-SA | Oral Nicotine 24
Number analyzed (Participants) | 36 | 34
(ng/ml) | 4.49 (1.60) | 4.76 (1.45)

6. Primary Outcome: Average Concentration
Description: Pharmacokinetic measurement - average concentration during the last dosing interval (AUCtau)
Time Frame: During the last dosing interval (hour 11-12 post-dose)
Population: ITT
Measure: Geometric Mean (Standard Deviation); unit: (ng/ml)
Arm/Group | Oral Nicotine 24-SA | Oral Nicotine 24 | Oral Nicotine 48 | NiQuitin™ Lozenge 4 mg | Nicorette® Gum 4 mg
Number analyzed (Participants) | 39 | 35 | 32 | 35 | 32
(ng/ml) | 13.33 (5.55) | 14.04 (4.50) | 27.50 (9.18) | 23.70 (9.86) | 22.15 (7.49)

ADVERSE EVENTS:
Arm/Group | Oral Nicotine 24-SA | Oral Nicotine 24 | Oral Nicotine 48 | NiQuitin™ Lozenge 4 mg | Nicorette® Gum 4 mg
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/37 | 0/36 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 29/40 | 22/37 | 27/36 | 24/35 | 18/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Nicotine 24-SA (N=40) | Oral Nicotine 24 (N=37) | Oral Nicotine 48 (N=36) | NiQuitin™ Lozenge 4 mg (N=35) | Nicorette® Gum 4 mg (N=35)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 7 | 0 | 5 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 4 | 7 | 6 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 3 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Eructation (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 6 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Nausea (Gastrointestinal disorders) | 5 | 3 | 4 | 4 | 4 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Salivary hypersecretion (Gastrointestinal disorders) | 7 | 0 | 1 | 0 | 3 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3 | 3 | 0 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Headache (Nervous system disorders) | 10 | 6 | 10 | 7 | 7 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Hiccups (Respiratory, thoracic and mediastinal disorders) | 18 | 18 | 18 | 9 | 6 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 3 — Total number of subjects affected in the safety analysis set in arms where the data lies above the 5% threshold
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 3
Lacrimation Increase (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Diarrheoa (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Glossodynia (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0
Oropharyngial Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes